CLINICAL TRIAL: NCT02479906
Title: A Prospective, Double Blind, Randomized, Controlled Study to Evaluate the Safety and Efficacy of the Brainsway (HAC-Coil) Deep Transcranial Magnetic Stimulation (DTMS) System for the Treatment of Post-Traumatic Stress Disorder (PTSD)
Brief Title: A Safety & Efficacy Study With Deep Transcranial Magnetic Stimulation for the Treatment of Post-Traumatic Stress Disorder (PTSD)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The results did not demonstrate sufficient clinical benefit induced specifically by the active treatment to justify continuation of the trial.
Sponsor: Brainsway (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTP-PTSD-01
Record Dates: First submitted 2015-06-15; First posted 2015-06-24 (Estimated); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Post-Traumatic Stress Disorder; PTSD; dTMS
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham Treatment (Sham Comparator): In the sham treatment,the electrical field induced by the sham coil cannot invoke any action potentials and if no action potentials are induced, then the electric field is insignificant and there is no treatment effect on the brain.
  Interventions: Device: Sham Treatment
- Deep TMS System (Experimental): Deep Transcranial Magnetic Stimulation (DTMS) is a new form of TMS which allows direct stimulation of deeper neuronal pathways than the standard TMS. The HAC Coil is designed to stimulate neuronal pathways in the medial prefrontal cortex or motor cortex, including the anterior cingulated cortex.
  Interventions: Device: Deep TMS System

INTERVENTIONS:
Device: Deep TMS System — Deep TMS treatments will be administered 3 times a week for 4 weeks and additional 2 booster treatments at the 5 and 9 week follow-up visits, for a total of 14 treatment sessions.
  Arms: Deep TMS System
Device: Sham Treatment — Sham treatments will be administered 3 times a week for 4 weeks and additional 2 booster treatments at the 5 and 9 week follow-up visits, for a total of 14 treatment sessions
  Arms: Sham Treatment

SUMMARY:
The purpose of the present study is to evaluate the safety and efficacy of Brainsway Deep TMS (DTMS) for the treatment of PTSD.

DETAILED DESCRIPTION:
Deep TMS in conjunction with brief trauma exposure will be compared to sham treatment in conjunction with brief trauma exposure, in a multicenter, randomized, controlled study for the treatment of PTSD. Study duration is 9 weeks, consisting of 4 weeks of treatment and a 5 week and 9 week follow-up visit. Subjects will be randomized to real or sham treatment stratified by site. The design is meant to demonstrate that the device shows superiority compared to sham treatment at the 5 week follow-up visit and at the 9 week follow-up visit, 1 month post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* Men and women 22-68 years of age
* Subjects currently diagnosed with PTSD according to the DSM-5, using the CAPS-5 (past-month version), with the following criteria met:

  * Criterion B: at least 1/5 intrusion symptoms; and
  * Criteria C: at least 1/2 avoidance symptoms; and
  * Criteria D: at least 2/7 cognition & mood symptoms; and
  * Criteria E: at least 2/6 arousal & reactivity symptoms; and
  * Criterion F: duration is met; and
  * Criteria G: distress is met.
* Subjects with at least moderate PTSD with a CAPS-5 score ≥ 25 at both Screening and Baseline visits.
* Subjects with an HDRS-21 score ≤ 26 at both Screening and Baseline visits.
* Subjects with negative or mitigated answers on safety screening questionnaire for transcranial magnetic stimulation.
* Negative pregnancy test in childbearing age women.
* Subject is capable and willing to provide informed consent.
* Subject is able to adhere to the treatment schedule.

Exclusion Criteria:

* Subject diagnosed according to the SCID I as suffering from any other major Axis I disorder, such as Psychotic Disorder, Bipolar affective disorder, OCD (MDD is not contraindicated when HDRS-21≤26).
* Subjects diagnosed according to the SCID II as suffering from Severe Personality Disorder.
* Subjects with significant suicidal risk as assessed by the investigator using the Beck Suicide Ideation scale, psychiatric interview or a history of attempted suicide in the past year.
* Subject has a history of epilepsy or seizure (EXCEPT those therapeutically induced by ECT).
* Subject has a history of significant head trauma with loss of consciousness for longer than 5 minutes.
* Subject has a history of cranial surgery.
* Subject has metallic particles in the eye or head (exclusive of mouth), implanted cardiac pacemaker or any intra-cardiac lines, implanted neurostimulators, intra-cranial implants (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or implanted medical pumps.
* Subject has severe and frequent headaches.
* Subject has a history of significant hearing loss.
* Subjects with a significant neurological disorder or insult including, but not limited to:

  * Any condition likely to be associated with increased intracranial pressure
  * Space occupying brain lesion
  * History of cerebrovascular accident
  * Transient ischemic attack within two years
  * Cerebral aneurysm
  * MMSE ≤ 24
  * Parkinson's disease
  * Huntington's chorea
  * Multiple sclerosis
* Subject with a history of substance abuse including alcoholism within the past 6 months (except nicotine and caffeine).
* Inadequate communication with the patient.
* Subject is under custodial care.
* Subject is currently participating in another clinical study or enrolled in another clinical study within 30 days prior to this study.
* Subject with unstable physical disease such as unstable cardiac disease.
* Subject is currently on Benzodiazepine at a dose higher than 3 mg of Lorazepam or equivalent.
* Subject has had previous treatment with TMS.
* Women who are breast-feeding.
* Women of childbearing potential and not using a medically accepted form of contraception when sexually active.

Ages: 22 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2016-11-17 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
CAPS-5 Score | 5 weeks from baseline
  CAPS-5 Score measured by change from baseline.

SECONDARY OUTCOMES:
Response Rate | 5 weeks from baseline
  Response rate at the 5 week follow-up visit.

OTHER OUTCOMES:
Adverse events | 5 and 9 weeks
  Measured by vital signs, physical & neurological examinations, lack of significant increase in suicide ideation, & other adverse event reporting.
Changes in Cognitive Scales | 5 and 9 weeks
  Changes in MMSE and BSRT Scales

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Isserles, MD, Principal Investigator — Hadassah Ein Karem Medical Center and Center for Addiction and Mental Health (CAMH); Zafiris J. Daskalakis, MD, Principal Investigator — Center for Addiction and Mental Health (CAMH); Avraham Zangen, PhD, Principal Investigator — Ben-Gurion University of the Negev
Locations (15):
- United States (12):
  - CalNeuro Research Group, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California - San Diego Medical Center, San Diego, California
  - Kadima Neuropsychiatry, San Diego, California
  - University of Florida College of Medicine, Gainesville, Florida
  - Advanced Mental Health Care Inc. - Juno Beach, Juno Beach, Florida
  - Advanced Mental Health Care Inc.-Palm Beach, Palm Beach, Florida
  - Advanced Mental Health Care Inc. - Royal Palm Beach, Royal Palm Beach, Florida
  - Yellowbrick Foundation, Evanston, Illinois
  - TMS Hope Center of Long Island, New York, New York
  - Carolina Partners in Mental Healthcare PLLC, Raleigh, North Carolina
  - Medical University Of South Carolina (MUSC), Charleston, South Carolina
- Center for Addiction and Mental Health (CAMH), Toronto, Ontario, Canada
- Israel (2):
  - Be'er Yaacov Mental Health Center, Be’er Ya‘aqov
  - Tel Hashomer Hospital, Tel Litwinsky

REFERENCES:
- [Derived] Isserles M, Tendler A, Roth Y, Bystritsky A, Blumberger DM, Ward H, Feifel D, Viner L, Duffy W, Zohar J, Keller CJ, Bhati MT, Etkin A, George MS, Filipcic I, Lapidus K, Casuto L, Vaishnavi S, Stein A, Deutsch L, Deutsch F, Morales O, Daskalakis ZJ, Zangen A, Ressler KJ. Deep Transcranial Magnetic Stimulation Combined With Brief Exposure for Posttraumatic Stress Disorder: A Prospective Multisite Randomized Trial. Biol Psychiatry. 2021 Nov 15;90(10):721-728. doi: 10.1016/j.biopsych.2021.04.019. Epub 2021 May 4. PMID 34274108